CLINICAL TRIAL: NCT00678938
Title: General Population Based Interventions for Smokers Not Ready to Quit: Testing Smoking Reduction vs. Abstinence Oriented Computer Expert Systems
Brief Title: Smoking Interventions in the General Population
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Christian Meyer, Dr. (principal investigator) / Anja Schumann, Dr. (co-investigator) / Ulrich John, Prof. Dr. (study director), Ernst-Moritz-Arndt-University of Greifswald, Institute of Epidemiology and Social Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: E2_P5, 01EB0420
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Tobacco Smoking
Keywords: smoking reduction; smoking cessation; stages of change; expert system interventions
MeSH Terms: conditions — Tobacco Smoking; Smoking Reduction; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Smoking abstinence oriented expert system intervention
- 2 (Experimental)
  Interventions: Behavioral: Smoking reduction oriented expert system intervention
- 3 (No Intervention)

INTERVENTIONS:
Behavioral: Smoking abstinence oriented expert system intervention — Participants received up to three counselling letters targeting smoking cessation
  Arms: 1
Behavioral: Smoking reduction oriented expert system intervention — Participants received up to three counselling letters targeting smoking reduction
  Arms: 2

SUMMARY:
The study takes up two problems: 1) Little research exists about general population interventions for smokers not ready to quit within the foreseeable future. 2) There is little evidence for smoking reduction as a behavioural goal in interventions. Interventions based on the Transtheoretical Model of Behavior Change (TTM) using computer expert-system technology yield delayed and smaller effects in smokers in the precontemplation stage of change compared to smokers in more advanced stages of change. Reducing the number of cigarettes smoked per day is currently discussed as an intermediate goal for this subgroup. Epidemiological and clinical studies revealed that smokers are able to maintain a substantial reduction. No undermining effects with respect to smoking cessation have been found. However, there are no studies that test the efficacy of behavioural interventions for smoking reduction using population based recruitment. Objectives: Testing the efficacy of TTM based interventions for general population smokers not intending to quit smoking, i.e. a smoking-reduction and a smoking-cessation tailored intervention using computerized expert-system technology.

ELIGIBILITY:
Inclusion Criteria:

* Daily smoking of 10 or more cigarettes
* No intention to quit within the next six month
* Age of 18 years and older
* valid telephone number

Exclusion Criteria:

- Insufficient german language and cognitive capabilities to complete the assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1462 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Point prevalence of tobacco abstinence | 24 hours, 7 days, 4 weeks, 6 months preceeding the 12 and 24 month follow-up assessments

SECONDARY OUTCOMES:
number of Cigarettes smoked per day | 4 weeks preceeding follow-up assessment
number of quit and cutdown attempts | last 12 months preceeding follow-up assessment
Stages of change progress | at 12 and 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, Dr., Principal Investigator — Ernst-Moritz-Arndt-University of Greifswald, Institute of Epidemiology and Social Medicine; Ulrich John, Prof. Dr., Study Director — Ernst-Moritz-Arndt-University of Greifswald, Institute of Epidemiology and Social Medicine